CLINICAL TRIAL: NCT06127069
Title: Treatment of Residual Pockets in Periodontal Patients Using an Oscillating Chitosan Device - A Randomized Parallel Arm Clinical Trial
Brief Title: Treatment of Residual Pockets in Periodontal Patients Using an Oscillating Chitosan Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgia Tseleki, Postgraduate Student, principal investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14/07/2021, 129
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis
Keywords: residual pockets; chitosan; treatment of periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: randomized parallel arm clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chitosan group (Experimental): debridement of residual periodontal pockets with ultrasonic scaler and the chitosan brush
  Interventions: Device: chitosan brush; Device: ultrasonic scaler
- control group (Active Comparator): debridement of residual periodontal pockets with ultrasonic scaler only
  Interventions: Device: ultrasonic scaler

INTERVENTIONS:
Device: chitosan brush — debridement of periodontal pockets with ultrasonic scaler first and after with chitosan brush for 2 minutes
  Other Names: Labrida BioClean
  Arms: chitosan group
Device: ultrasonic scaler — debridement of periodontal pockets only with ultrasonic scaler

SUMMARY:
The aim of the current study was to investigate the effect of a chitosan brush on the treatment of residual pockets in patients already treated for periodontal disease. Thirty-six patients with chronic periodontitis (Stage ΙΙΙ, ΙV) that had already completed causative therapy and exhibited at least two residual periodontal pockets ≥ 5mm that bled on probing, were randomly assigned to two groups. In the test group debridement of residual pockets was performed with ultrasonic scaler and the chitosan brush, whereas in the control group only ultrasonic scalers were used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 or over
* Subjects diagnosed with chronic periodontitis, Stage III or IV, and had received full mouth scaling and root planning at least three months prior to baseline examination
* Subjects with at least two residual periodontal pockets of at least 5mm depth that bled on probing
* Full mouth plaques scores ≤20%

Exclusion Criteria:

* Subjects that had received antibiotic therapy 6 months prior to initial examination
* Subjects with compromised systemic conditions
* Patients undergoing chemotherapy or radiotherapy
* Pregnant or lactating women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-11-29 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth | baseline, 6 weeks, 3 months, 6 months
  the distance from the mucosa margin to the bottom of the periodontal pocket
MMP-8 | baseline, 6 weeks, 3 months, 6 months
  levels of matrix metalloproteinase -8 in gingival crevicular fluid

SECONDARY OUTCOMES:
Bleeding on Probing | baseline, 6 weeks, 3 months, 6 months
  presence or absence of bleeding after probe insertion in the periodontal pocket
Clinical Attachment Level | baseline, 6 weeks, 3 months, 6 months
  the distance from cementoenamel junction to the bottom of periodontal pocket
Gingival Recession | baseline, 6 weeks, 3 months, 6 months
  the distance from cementoenamel junction to the mucosa margin

CONTACTS AND LOCATIONS:
Overall Officials: Lazaros Tsalikis, Study Chair — Department of Periodontology, School of Dentistry, Aristotle University
Locations (1):
- Department of Periodontology, School of Dentistry, Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tseleki G, Batas L, Davidopoulou S, Wohlfahrt JC, Menexes G, Tsalikis L. Management of residual periodontal pockets using an oscillating chitosan device: A randomized clinical trial. J Periodontol. 2025 Nov 7. doi: 10.1002/jper.70010. Online ahead of print. PMID 41201882